CLINICAL TRIAL: NCT01310179
Title: Phase I, Open-label Study Evaluating the Safety of Escalating Doses of Ad/PNP-F-araAMP (Ad/PNP Administered Intratumorally With Co-administration of Fludarabine Phosphate Intravenously) in Subjects With Advanced Solid Tumors
Brief Title: Safety Study of Adenovirus/PNP Coupled With Fludarabine Phosphate to Treat Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PNP Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNP-001
Record Dates: First submitted 2011-03-03; First posted 2011-03-08 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer
Keywords: gene therapy; advanced solid tumors; Head and Neck cancer; intratumoral therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad/PNP and fludarabine monophosphate (Experimental): Ad/PNP will be injected three times into the tumor over 2 days followed by three daily intravenous infusions of F-araAMP (fludarabine monophosphate). Subjects in the first 3 cohorts will receive 3x10e11 VP for 3 injections and escalating dose levels of F-araAMP (15, 45, and 75 mg/m2 in each sequential cohort) daily for 3 days. The fourth cohort will receive 3x10e12 for 3 injections and 75 mg/m2 fludarabine daily for 3 days.
  Interventions: Genetic: Ad/PNP and fludarabine monophosphate

INTERVENTIONS:
Genetic: Ad/PNP and fludarabine monophosphate — Subjects in the first 3 cohorts will receive 3x10e11 VP for 3 injections and escalating dose levels of F-araAMP (15, 45, and 75 mg/m2 in each sequential cohort) daily for 3 days. The fourth cohort will receive 3x10e12 for 3 injections and 75 mg/m2 fludarabine daily for 3 days.

SUMMARY:
This study will test whether it is possible to introduce new genetic material into a small portion of a tumor and have the product of the new gene not only kill those tumor cells that were infected initially, but also the surrounding tumor cells as well with limited or no harm to the patient. The desired effects of this approach are achieved by focusing potent chemotherapies directly within the tumor itself and, as a result, avoiding injury to the remainder of the body. In this study, we will use two components, the first of which is a virus, known as an adenovirus, that has been crippled (i.e., it cannot make more of itself) and loaded with a bacterial gene called E. coli purine nucleoside phosphorylase (PNP). Adenoviruses are considered to be relatively safe vehicles for gene delivery and are presently being used in numerous human trials and therapies worldwide, including a head and neck cancer therapy approved for use outside the United States. The loaded adenovirus will be used to deliver the PNP gene directly into a tumor in patients. This gene is not expected to have an effect itself. However, the gene produces PNP inside the tumor and this protein will activate the second component of the therapy, a drug called fludarabine phosphate, which is approved by the FDA for certain types of blood-cell cancers, but has not been shown to be effective against most solid tumors. The proposed therapy gives the patient several infusions of fludarabine following the injection of the virus carrying the PNP gene and, as the fludarabine enters the tumor, it will be converted by PNP into a second compound, fluoroadenine. Numerous studies in mice and rats have shown that fluoroadenine is a very potent anti-cancer agent and that it will kill the tumor cells where it is made as well as those in the immediately surrounding area.

DETAILED DESCRIPTION:
For this first study, we will inject the PNP-loaded adenovirus into the tumors of patients with cancers primarily in the throat and neck and then give them the drug. This study is designed with two goals in mind: 1) assessing the overall safety of this approach for the patient; and 2) observing the effects of this anti-cancer strategy on the tumor itself. This will be accomplished in two parts. First, we will introduce a modest, fixed amount of the gene-carrying adenovirus into the tumors of three separate groups of patients and then administer small, increasingly strong amounts of the fludarabine phosphate to each successive group over a three-day period. Even in the group that will receive the highest amount of fludarabine, the total amount given to any individual patient over those three days will be significantly less than the dose approved by the FDA for patients with non-solid tumors. Finally, a more concentrated amount of the adenovirus (approximately 10 times more viruses) will be given to a fourth group of patients who will also receive the highest dose of the drug that was shown to be well tolerated in the prior three groups (the highest dose at which no serious problems were observed).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of a solid tumor
* Failed or exhausted all standard or approved treatment options that would provide substantive palliation
* Have at least one measurable primary or metastatic tumor on imaging studies or physical exam whose potential reduction could provide relief of symptoms or benefit
* Tumor is accessible for direct intratumoral injection

Exclusion Criteria:

* Diagnosis of leukemia
* Have previously received any gene therapy products or oncolytic viral therapy
* Receiving treatment with allopurinol
* Received radiation treatment < 4 wks prior to first injection of Ad/PNP
* Received chemotherapy < 4 wks prior to first injection of Ad/PNP
* Have signs or symptoms of active infection
* Receiving chronic systemic corticosteroids or any chronic immunosuppressive medications within 14 days prior to first injection of Ad/PNP. Subjects receiving short courses of corticosteroids are considered eligible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Rosenthal EL, Chung TK, Parker WB, Allan PW, Clemons L, Lowman D, Hong J, Hunt FR, Richman J, Conry RM, Mannion K, Carroll WR, Nabell L, Sorscher EJ. Phase I dose-escalating trial of Escherichia coli purine nucleoside phosphorylase and fludarabine gene therapy for advanced solid tumors. Ann Oncol. 2015 Jul;26(7):1481-7. doi: 10.1093/annonc/mdv196. Epub 2015 Apr 21. PMID 25899782

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ad/PNP and Fludarabine Monophosphate
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ad/PNP and Fludarabine Monophosphate
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance Status Score [Number; unit: participants] — The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death. The primary purpose of its development was to allow physicians to evaluate a patient's ability to survive chemotherapy for cancer.
  100 - Normal; no complaints; no evidence of disease.
  90 - Able to carry on normal activity; minor signs or symptoms of disease.
  80 - Normal activity with effort; some signs or symptoms of disease.
  70 - Cares for self; unable to carry on normal activity or to do active work.
  participants
    100% | 2
    90% | 3
    80% | 3
    70% | 4
Tumor Site [Number; unit: participants] — location of primary tumor
  participants
    Neck | 6
    Cheek | 1
    Hard Palate | 1
    Tonsil | 1
    Lower Lip | 1
    Scalp | 1
    Lower Extremities | 1
Tumor Histology [Number; unit: participants]
  squamous cell carcinoma | 8
  adenoid cycstic carcinoma | 2
  melanoma | 2
Recurrence [Number; unit: participants]
  Local | 7
  Regional | 4
  Distant | 1
Non-Target Lesions [Number; unit: participants] — presence or absence of additional cancerous lesions that were not treated with the study drug
  participants
    Present | 7
    Not Present | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Effects After Ad/PNP-F-araAMP Treatment
Description: Number of participants who had the most frequently observed undesirable effects after exposure to study drug
Time Frame: Entry through Study Day 56
Measure: Number; unit: participants
Groups:
- Ad/PNP and Fludarabine Monophosphate: Ad/PNP will be injected three times into the tumor over 2 days followed by three daily intravenous infusions of F-araAMP (fludarabine monophosphate). Subjects in the first three cohorts will receive 3x10e11 VP for 3 injections and 5, 15 or 25 mg/m2 of F-araAMP daily for 3 days. Subject in the fourth cohort will receive 3x10e12 VP for 3 injections and the highest tolerated dose of F-araAMP daily for 3 days.
  Ad/PNP and fludarabine monophosphate: Subjects in the first 3 cohorts will receive 3x10e11 VP for 3 injections and escalating dose levels of F-araAMP (15, 45, and 75 mg/m2 in each sequential cohort) daily for 3 days. The fourth cohort will receive 3x10e12 for 3 injections and 75 mg/m2 fludarabine daily for 3 days.
Arm/Group | Ad/PNP and Fludarabine Monophosphate
Number analyzed (Participants) | 12
participants
  injection site symptoms | 12
  fatigue | 8
  facial pain | 8
  nausea | 5

2. Secondary Outcome: Treatment Outcome and Percent Change in Tumor Volume
Description: Measurement of tumor response to study drug, as measured by the percentage of change in tumor volume as measured by a physicial measurement using a ruler
Time Frame: Entry through Study Day 56
Measure: Number; unit: participants
Arm/Group | Ad/PNP and Fludarabine Monophosphate
Number analyzed (Participants) | 12
participants
  Progression (>+20%) | 2
  Stable (+20% to -30%) | 5
  Partial Response (>-30%) | 5

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Ad/PNP and Fludarabine Monophosphate
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ad/PNP and Fludarabine Monophosphate (N=12)
dehydration (Metabolism and nutrition disorders) | 1
pericardial effusion (Cardiac disorders) | 1
cardiac tamponade (Cardiac disorders) | 1
pain (General disorders) | 1
nausea/vomiting (Gastrointestinal disorders) | 1
bacteremia (Infections and infestations) | 1
partial seizure (Nervous system disorders) | 1
lower extremity weakness (Musculoskeletal and connective tissue disorders) | 1
chronic wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ad/PNP and Fludarabine Monophosphate (N=12)
injection site symptoms (General disorders) | 12
fatigue (General disorders) | 8
facial pain (General disorders) | 8
nausea (Gastrointestinal disorders) | 5
flu-like symptoms (General disorders) | 4
dizziness (Nervous system disorders) | 4
headache (Nervous system disorders) | 4
decreased lymphocytes (Metabolism and nutrition disorders) | 4
decreased hemoglobin (Metabolism and nutrition disorders) | 4
decreased/loss of appetite (Metabolism and nutrition disorders) | 4
paresthesia (Nervous system disorders) | 4
non-cardiac chest pain (General disorders) | 3
facial edema (General disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 3
hypertension (Vascular disorders) | 3
yeast infection (Infections and infestations) | 3
sore throat (Respiratory, thoracic and mediastinal disorders) | 3
back pain (Musculoskeletal and connective tissue disorders) | 2
lower extremity edema (General disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 2
pruritis (Skin and subcutaneous tissue disorders) | 2
neck stiffness (Musculoskeletal and connective tissue disorders) | 2
dysphagia (Gastrointestinal disorders) | 2
tachycardia (Cardiac disorders) | 2
hypotension (Vascular disorders) | 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
constipation (Gastrointestinal disorders) | 2
syncope (Nervous system disorders) | 2
arm pain (Musculoskeletal and connective tissue disorders) | 1
vomiting (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
increased AST (Metabolism and nutrition disorders) | 1
fever (General disorders) | 1
urinary urgency (Renal and urinary disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
chills (General disorders) | 1
hypothyroidism (Endocrine disorders) | 1
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
pericardial effusion (Cardiac disorders) | 1
upper respiratory infection (Infections and infestations) | 1
localized edema (General disorders) | 1
periorbital edema (Skin and subcutaneous tissue disorders) | 1
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
wound infection (Infections and infestations) | 1
dehydration (Metabolism and nutrition disorders) | 1
wheezing (Respiratory, thoracic and mediastinal disorders) | 1
acute renal failure (Renal and urinary disorders) | 1
oral mucositis (Gastrointestinal disorders) | 1
weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No